CLINICAL TRIAL: NCT00780702
Title: Aripiprazole for Prevention of Relapse to Cocaine Use in Methadone-Maintenance Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999908426; 08-DA-N426
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-02-27

CONDITIONS: Cocaine Dependence; Cocaine-Related Disorders; Opioid-Related Disorders
Keywords: Cocaine; Treatment; Airpiprazole; Methadone; Relapse; HIV; Ecological Momentary Assessment (EMA); Contingency Management
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Recurrence

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Airipiprazole
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Airipiprazole — Participants receive aripiprazole (orally, up to 15 mg/day) plus standard methadone maintenance (daily oral methadone and weekly individual counseling).
  Arms: Arm 1
Drug: Placebo — Participants receive identical capsules containing no active medication plus standard methadone maintenance (daily oral methadone and weekly individual counseling).
  Arms: Arm 2

SUMMARY:
Background:

* The effectiveness of methadone maintenance for treatment of heroin addiction has been well established. However, patients maintained on methadone may relapse to cocaine use, even when they are enrolled in a comprehensive treatment program. Relapse has been attributed to several factors, including drug-associated environmental stimuli.
* Aripiprazole is a drug used to treat schizophrenia and bipolar disorder, but it may have other uses. Research has shown that aripiprazole can reduce cocaine-seeking behavior in rats, and it has been investigated for use in treating amphetamine dependence. More research is needed to determine whether aripiprazole can prevent relapse to cocaine use in patients being treated with methadone.

Objectives:

- To determine whether aripiprazole prevents relapse to cocaine use more effectively than placebo in cocaine-abstinent patients maintained on methadone.

Eligibility:

- Individuals between 18 and 60 years of age who are current cocaine users seeking methadone treatment.

Design:

* The study will last up to 41 weeks, with four phases of treatment and a follow-up evaluation. Three times a week, participants will be asked to report illicit drug use and provide urine and breath samples. Throughout the study, participants will receive individual counseling in weekly 40 60 minute sessions. Other samples and tests will be scheduled as required by the study researchers.
* Patients will be stabilized on daily methadone over the first 14 days of the study.
* Weeks 1 14: Participants will receive vouchers for regular cocaine-free urine samples. Those who successfully complete this phase will continue to the next part of the study.
* Weeks 13 27: Participants will receive either aripiprazole or placebo along with their methadone. During this part of the study, participants will keep electronic diaries to record cocaine use or craving and to record data on mood and activity.
* Weeks 28 33: Participants will stop taking the aripiprazole or placebo, but will continue the methadone treatment. Participants will continue to use the electronic diaries.
* Weeks 34 41: Participants will have the choice of transferring to a community clinic or gradually reducing doses of methadone to end the study.
* Participants will return for a follow-up visit and urine sample 6 months after the end of the study.

DETAILED DESCRIPTION:
Background. Though methadone effectively treats opioid dependence in polydrug users, some abstinent patients relapse to maladaptive use of cocaine during treatment. Relapse may be triggered by cocaine-associated cues. Work in a rodent relapse model has demonstrated that the atypical neuroleptic drug aripiprazole (Abilify), a partial agonist at dopamine D2 receptors, can block relapse to cocaine use induced by cocaine-associated environmental stimuli or by priming doses of cocaine.

Scientific goals. To determine whether aripiprazole prevents relapse to cocaine use more effectively than placebo in cocaine-abstinent patients maintained on methadone.

Participant population. A total of up to 275 opioid-dependent outpatients abusing cocaine and opioids (110 evaluable) will be enrolled. Target enrollment will include 40% women and 60% minorities (mostly African-American).

Experimental design and methods. The study will be a randomized double-blind clinical trial with two treatment groups (55 per group): aripiprazole (15 mg oral daily) and placebo. All patients will receive standard treatment (methadone daily and individual counseling weekly) for 39 weeks. To establish abstinence prior to aripiprazole induction, contingent vouchers will be given for each cocaine-negative urine specimen during the first 12 weeks (weeks 1-12). Participants who are abstinent from cocaine during weeks 11 and 12 will be randomized to receive aripiprazole or aripiprazole placebo in weeks 13 through 27 (induction, weeks 13 and 14; taper, week 27). From weeks 28-33, participants will receive methadone and counseling only, and then will be offered assistance to transfer to another program; those who do not transfer will undergo an 8-week methadone detoxification. The primary outcome measures will be time to relapse and longest duration of cocaine abstinence. Secondary objectives include evaluating whether the treatment groups differ in self-reported changes in drug use and proportion of drug-negative urine specimens. In addition, drug use, drug craving, stress, and HIV-risk behaviors such as injection practices will be assessed via electronic diaries (ecological momentary assessment, EMA).

Benefits to participants and/or society. Participants will receive methadone, drug counseling, and contingency-management therapy. The methadone, counseling, and voucher interventions are likely to reduce participants use of heroin and cocaine and HIV risk behaviors. Aripiprazole may reduce the incidence of relapse to cocaine use.

Risks to participants. Participants may experience side effects from aripiprazole and methadone and discomfort during withdrawal from methadone and aripiprazole. Methadone could raise serum levels of aripiprazole via inhibition of CYP2D6 metabolic pathways. The EMA component of the study may generate some assessment burden.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18 and 60
  2. Evidence of physical dependence on opioids (determined by self-report, urine screen, and physical exam)
  3. Evidence of (a) current cocaine use (determined by self-report and urine screen) or (b) cocaine dependence (DIS interview for DSM-IV criteria).
  4. Lifetime drug-use duration of at least 1 year and current cocaine use on at least 3 days of the last 30.
  5. Seeking treatment for opiate and cocaine use.
  6. Able to attend methadone clinic 7 days/week.

EXCLUSION CRITERIA:

1. Any medical illness that in the view of the investigators would compromise participation in research (determined by Self-Reported Medical History; Physical Examination; Blood and Urine Laboratory tests; see details under Screening measures below), including, but not limited to:

   * cardiovascular disease
   * cerebrovascular disease
   * unexplained history of syncope
   * history of seizures, except for febrile seizures at childhood
   * chronic renal failure, as estimated by Cr > 2.0
   * diabetes mellitus
   * hyperlipidemia
2. Allergy, hypersensitivity, or intolerance to either methadone or aripiprazole (determined by Self-Reported Medical History)
3. AIDS, CD4 <200, or evidence of severely compromised immune system (determined by Blood Laboratory tests; see details under Screening measures below)
4. Pregnancy or breastfeeding (Urine Pregnancy Test; self report)
5. Orthostatic hypotension (i.e., upon standing for 3 minutes, a 20 mm Hg decrease in systolic blood pressure or a 10 mmHg decrease in diastolic blood pressure, accompanied by an increase by 20 bpm in heart rate) on two separate readings during physical examination.
6. Marked, sustained high blood pressure (SBP >160 mm Hg, DBP >100 mm Hg) on two or more readings at a single visit and confirmed with two readings on a follow-up visit. If a participant is started on antihypertensive drugs at the start of the study, the participant may be cleared, but will not be started on aripiprazole until confirmation that the hypertension is well controlled (systolic blood pressure < 150, diastolic blood pressure < 100 mm Hg) on two readings at least 3 days apart.
7. ECG abnormalities including QTc interval > 450 ms or changes suggesting acute ischemia, <TAB>second or third degree heart block, left bundle branch block, atrial fibrillation, or other <TAB>clinically important arrhythmias. ECGs may be sent to an outside cardiologist for manual <TAB>reading.
8. Contraindicated medications (Self-Reported Medical History):

   * Alpha-1 receptor blockers (e.g., doxazin, terazosin)
   * Anti-epileptic medications (e.g., carbamazepine)
   * Tricyclic antidepressants
   * SSRIs
   * Neuroleptics
   * Quinidine
   * Antifungals (e.g., ketoconazole)
   * Ranolazine
   * CYP3A4 inhibitors or inducers (other than methadone)
   * CYP2D6 inhibitors or inducers (other than methadone)
9. Family history (Self-Reported Medical History):

   * Family history of sudden death of unexplained causes
   * Sudden cardiac death
   * Aneurysm
   * Myocardial infarction below the age 50 years
10. Psychiatric history:

    A) Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires (Shipley Institute of Living scale estimated full-scale IQ less than 80)

    B) History of schizophrenia or any other DSM-IV psychotic disorder (Self-Reported Medical History; Diagnostic Interview Schedule for the DSM-IV (DIS IV))

    C) History of bipolar disorder (Self-Reported Medical History; DIS IV)

    D) Current Major Depressive Disorder (Self-Reported Medical History; DIS IV)

    E) Previous suicide attempts or ideation (Self-Reported Medical History; DIS-IV)

    F) Dementia (DIS-IV; Clinical Interview; Shipley Institute of Living scale)
11. Current physical dependence on alcohol or sedative-hypnotics, e.g. benzodiazepines (self-report; ASI; alcohol CAGE questions; and pattern of positive drug screens or BAL for alcohol)
12. Body Mass Index (BMI) over 40
13. Failure to agree to use a medically effective form of contraception while in the study (in women who are sexually active with a male partner and able to get pregnant). Acceptable forms of contraception for this study include:

    * hormonal contraceptives (birth control pills, injectable hormones, vaginal ring hormones),
    * surgical sterility (tubal ligation or hysterectomy)
    * IUD
    * Diaphragm with spermicide
    * Condom with spermicide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2008-05-08; Primary Completion 2013-04-16 (Actual); Study Completion 2013-04-16 (Actual)

PRIMARY OUTCOMES:
Time to relapse | 19 weeks

SECONDARY OUTCOMES:
Cocaine use | 19 weeks
HIV risk behaviors | 19 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bjornsson TD, Callaghan JT, Einolf HJ, Fischer V, Gan L, Grimm S, Kao J, King SP, Miwa G, Ni L, Kumar G, McLeod J, Obach SR, Roberts S, Roe A, Shah A, Snikeris F, Sullivan JT, Tweedie D, Vega JM, Walsh J, Wrighton SA; Pharmaceutical Research and Manufacturers of America Drug Metabolism/Clinical Pharmacology Technical Working Groups. The conduct of in vitro and in vivo drug-drug interaction studies: a PhRMA perspective. J Clin Pharmacol. 2003 May;43(5):443-69. PMID 12751267
- [Background] Childress AR, O'Brien CP. Dopamine receptor partial agonists could address the duality of cocaine craving. Trends Pharmacol Sci. 2000 Jan;21(1):6-9. doi: 10.1016/s0165-6147(99)01422-4. No abstract available. PMID 10637646
- [Background] Conley RR, Kelly DL, Gale EA. Olanzapine response in treatment-refractory schizophrenic patients with a history of substance abuse. Schizophr Res. 1998 Sep 7;33(1-2):95-101. doi: 10.1016/s0920-9964(98)00062-0. PMID 9783349